CLINICAL TRIAL: NCT00002847
Title: TREATMENT OF METASTATIC RENAL CELL CARCINOMA WITH SUBCUTANEOUS RECOMBINANT INTERLEUKIN-2 AND INTERFERON ALPHA
Brief Title: Interferon Alfa and Interleukin-2 in Treating Patients With Metastatic Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blumenthal Cancer Center at Carolinas Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065086; CMC-09-95-14B; NCI-V96-1039
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2003-12

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system to try to stop cancer cells from growing. Combining interferon alfa and interleukin-2 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of interferon alfa and interleukin-2 in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the response and disease-free survival of patients with metastatic renal cell carcinoma treated with subcutaneous interleukin-2 and interferon alfa.
* Assess the toxicity of this regimen.

OUTLINE: Patients undergo nephrectomy if the diseased kidney makes up the bulk of the tumor burden.

All patients receive subcutaneous interferon alfa on day 1 and interleukin-2 on days 3-5 of week 1, followed by reduced doses of interferon alfa and interleukin-2 on days 1, 3, and 5 of weeks 2-6. Patients are assessed for response approximately 2 months after initiating therapy. Patients with stable or responding disease undergo a second course; those who continue to respond may receive additional therapy provided toxicity is limited.

Patients are followed for survival.

PROJECTED ACCRUAL: 14 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven renal cell cancer that is metastatic

  * No greater than 50% estimated hepatic replacement by tumor on CT or MRI
  * No symptomatic involvement of the CNS or a major nerve
* Measurable disease required
* Ineligible for treatment with low-dose interleukin-2 on another CMC protocol

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50%-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* No coagulopathy (i.e., platelet count less than 80,000/mm3)

Hepatic:

* AST and ALT no greater than 5 times normal

Renal:

* Creatinine less than 4.0 mg/dL

Cardiovascular:

* No symptomatic angina
* No untreated coronary artery disease
* No refractory arrhythmia
* No abnormal left ventricular function

Pulmonary:

* No dyspnea on minimal exertion

Other:

* No site of ongoing bleeding
* No systemic infection
* No HIV antibody
* No HBsAg
* No requirement for steroids
* No psychiatric disease that precludes informed consent or protocol treatment
* No second malignancy except:

  * Basal cell skin carcinoma
  * Carcinoma in situ of the cervix
* Not pregnant or nursing
* Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interleukin-2

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 28 days since prior treatment for renal cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. White, MD, Study Chair — Blumenthal Cancer Center at Carolinas Medical Center
Locations (1):
- Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina, United States